CLINICAL TRIAL: NCT02634086
Title: Long-term Outcome of Triple-vessel Coronary Artery Disease Underwent Three Different Strategies (LOTUS)
Acronym: LOTUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Lei Song, MD, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: 2010CB732601
Record Dates: First submitted 2015-12-14; First posted 2015-12-17 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Coronary Artery Disease; Coronary Stenosis; Myocardial Ischemia
Keywords: Coronary artery disease; Percutaneous coronary intervention; Coronary artery bypass graft; Medication therapy
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Percutaneous coronary intervention: Patients with triple-vessel coronary artery disease underwent percutaneous coronary intervention.
- Coronary artery bypass graft: Patients with triple-vessel coronary artery disease underwent coronary artery bypass graft.
- Optimal medication therapy: Patients with triple-vessel coronary artery disease underwent optimal medication therapy only.

SUMMARY:
The study is to determine the long-term outcome of patients with coronary triple vessels disease (TVD) in the real world of China, by three different treatment strategies: percutaneous coronary intervention (PCI), Coronary artery bypass graft (CABG) or optimal medication therapy (OMT).

DETAILED DESCRIPTION:
About 10,000 participants will be enrolled into this retrospective study. Study coordinators will include both men and women over the age of 18 who had angiographic proved triple-vessel disease in a 15 years long-term. Detailed procedural data will be obtained by the study coordinator and local principal investigator. These data will be entered into the electronic data capture system. Participants will have telephone follow-up interviews conducted by the centralized follow-up center at Fuwai Hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has coronary angiography confirmed triple-vessel disease.
2. Subject is ≥ 18 years of age at the time of inclusion.
3. Subject is willing to comply with all protocol-required follow-up evaluation (patient will be followed during 1 month after hospital to assess any complications and clinical status).

Exclusion Criteria:

1. Subject is participating in another investigational clinical trial that may cause non-compliance with the protocol or confound data interpretation.
2. Female subjects with a positive quantitative or qualitative pregnancy test, in accordance with hospital policy.
3. Subjects with no way contact by telephone for follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between April 2004 and April 2018 in Fuwai Hospital, Beijing, China, consecutive patients with angiography confirmed triple-vessel coronary disease.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2004-04; Primary Completion 2016-04 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | Through study completion, an average of 5 year
  The mortality due to any cause

SECONDARY OUTCOMES:
Major adverse cardiac and cerebrovascular event | Through study completion, an average of 5 year
  The incidence rate of major adverse cardiac and cerebrovascular event (MACCE), which is a combination of all-cause death, myocardial infarction, stroke and repeat revascularization
Myocardial infarction | Through study completion, an average of 5 year
  The Incidence rate of myocardial infarction, including ST elevation myocardial infarction and non-ST elevation myocardial infarction
Stroke | Through study completion, an average of 5 year
  The incidence rate of stroke, including cerebral infarction and hemorrhage
Repeat revascularization | Through study completion, an average of 5 year
  The incidence rate of repeat revascularization, including target vessel revascularization and non-target vessel revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Lei Song, MD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Xu JJ, Zhang Y, Jiang L, Tian J, Song L, Gao Z, Feng XX, Zhao XY, Zhao YY, Wang D, Sun K, Xu LJ, Liu R, Gao RL, Xu B, Song L, Yuan JQ. Comparison of Long-term Outcomes in Patients with Premature Triple-vessel Coronary Disease Undergoing Three Different Treatment Strategies: A Prospective Cohort Study. Chin Med J (Engl). 2018 Jan 5;131(1):1-9. doi: 10.4103/0366-6999.221273. PMID 29271373